CLINICAL TRIAL: NCT00490334
Title: Assessment and Rehabilitation of Cognitive Impairments in Pediatric Survivors of Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-08123; 97817 (Other: Stanford University Alternate IRB Approval Number); PEDSVAR0003 (Other: OnCore)
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Neoplasms
Keywords: Carcinomas; Squamous Cel; Adenocarcinoma; Acute Lymphocytic Leukemia
MeSH Terms: conditions — Neoplasms; Carcinoma; Adenocarcinoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cancer patients: Children with cancer aged 8 to 16 years
- Control (non-cancer): Normal children aged 8 to 16 years, age- and gender-matched to the cancer cohort

SUMMARY:
This research involves assessment of cognitive outcome in childhood cancer as well as evaluation of a cognitive rehabilitation program for improving learning and problem solving difficulties in children with cancer.

DETAILED DESCRIPTION:
The purpose of this study is to help determine specific cognitive-behavioral and neurobiologic impairments associated with chemotherapy treatments in children with cancer and to assess the efficacy of a cognitive intervention program for improving cognitive impairments in these children.

ELIGIBILITY:
INCLUSION

Everyone:

* At least 9 years of age and less than 17 years

Patients

* Diagnosis of brain tumor or acute lymphocytic leukemia (ALL)
* Completed all anti-cancer treatment(s) including chemotherapy, radiation and/or surgery

Control group

* Typical for age

EXCLUSION

Everyone:

* Non-English speaking (translated cognitive testing and MRI assessments unavailable)
* MRI contraindication, including but not limited to orthodontia, metal implants, and/or pacemaker
* Major sensory deficit disorders, including but not limited to blindness or deafness

Patients

* Shunt placement
* Received bone marrow transplant
* History of neurologic, psychiatric, developmental or major medical condition (eg, diabetes) NOT related to cancer
* Participation in any concurrent cognitive rehabilitation study

Control group

* History of neurologic, psychiatric, developmental or major medical condition (eg, diabetes)

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric cancer patients 8 to 16 years of age, with age- and gender-matched control group.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2007-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Performance on neuropsychological testing and brain activation patterns measured by functional MRI | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shelli Kesler, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States